CLINICAL TRIAL: NCT03226821
Title: Body Composition and Adipose Tissue in HIV Lipodystrophy: Effects of Tesamorelin Therapy
Brief Title: Body Composition and Adipose Tissue in HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR2634; R01DK110771 (NIH)
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: HIV Lipodystrophy Syndrome; Growth Hormone Deficiency; Body Composition
Keywords: HIV Lipodystrophy; Tesamorelin; Body Composition; Visceral Adiposity
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Dwarfism, Pituitary | interventions — tesamorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tesamorelin (Experimental): Subjects will be treated with tesamorelin 2 mg by subcutaneous injection daily. Enrolled subjects will have 6 visits - a baseline visit before starting tesamorelin, a visit at 1 month, 3 months, 6 months, 9 months and at 1 year of tesamorelin (GHRH analogue) therapy. Blood sampling for safety labs and clinical examinations will be performed at each visit.
  Interventions: Drug: Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin — Patients will be treated with tesamorelin 2 mg by subcutaneous injection daily
  Other Names: Egrifta

SUMMARY:
In this study, the investigators will examine the effect of therapy with the Growth Hormone Releasing Hormone (GHRH) analog tesamorelin on body composition in patients with HIV lipodystrophy and central adiposity. This study is a single arm prospective study of tesamorelin therapy of patients with HIV lipodystrophy. Subjects will do body composition testing, adipose tissue biopsy, metabolic rate measurements and insulin sensitivity assessment before, 6 and 12 months after daily injections of tesamorelin 2 mg by subcutaneous injection.

DETAILED DESCRIPTION:
HIV lipodystrophy is increasingly recognized as a common and clinically significant long-term sequelae of HIV treatment. In the HIV lipodystrophy lipohypertrophy phenotype, visceral adipose tissue (VAT) is increased and this is associated with reduced growth hormone (GH) secretion. Mounting evidence also links this phenotype with dyslipidemia, insulin resistance, subclinical atherosclerosis and cardiovascular (CV) disease in patients with HIV disease. The etiology of HIV lipodystrophy (HIVLD) with central adiposity is unclear, but this phenotype is increasingly common with newer, less lipotoxic combination anti-retroviral therapy (cART) use. VAT and hepatic lipid accumulation, are important health concerns for HIVLD patients. This body composition pattern may contribute to the increased cardiovascular risk that has been demonstrated in patients with HIV lipodystrophy. Patients with HIVLD and central adiposity have been shown to have reduced GH secretion. Thus, a medication has been developed to augment GH secretion. This medication is tesamorelin. GH supplementation in other clinical settings has been shown to reduce visceral adiposity and may reduce hepatic lipid content.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected subjects with HIV lipodystrophy (HIVLD)
* Abdominal fat accumulation defined as: Waist Circumference (WC) 102 cm for men, 88 cm for women, except in subjects of East/South Asian ethnicity in whom this will be defined by WC 90 cm for men and 80 cm for women.
* Weight stable for 8 weeks prior to enrollment,
* CD4 count >100 cells/mm3
* HIV RNA load <1000 copies/mL
* Fasting plasma glucose <120 mg/dL
* Stable combination anti-retroviral therapy (cART) of any regimen for ≥ 8 weeks prior to study enrollment

Exclusion Criteria:

* Diabetes mellitus requiring medication
* History of any malignancy
* Abnormal renal or liver function
* Pregnancy or women of childbearing age who are not using an acceptable means of contraception
* History disorder of the hypothalamic-pituitary axis due to hypophysectomy, hypopituitarism or pituitary tumor/surgery
* Head irradiation or head trauma or adrenal insufficiency
* Systemic glucocorticoid use
* Known hypersensitivity to tesamorelin and/or mannitol

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Hepatic Lipid Content | Baseline and 12 months
  Hepatic lipid content measured by abdominal magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Change in Visceral Adipose Tissue (VAT) mass | Baseline and 12 months
  Visceral adipose tissue mass measured by abdominal MRI
Change in Relative gene expression of CD68 gene | Baseline and 12 months
  Relative gene expression of CD68 gene in adipose tissue
Change in Relative gene expression on TNF-alpha gene | Baseline and 12 months
  Relative gene expression of tumor necrosis factor (TNF)-alpha gene in adipose tissue
Change in Resting Energy Expenditure (REE) | Baseline and 12 months
  Resting metabolic rate measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U. Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit and Pituitary Center, Columbia University, New York, New York, United States